CLINICAL TRIAL: NCT01692795
Title: Cardiovascular Medication Prescriptions Before First Myocardial Infarction in Patients With and Without Previously Diagnosed Atherosclerotic Disease: an Analysis of Linked Prospectively Collected Electronic Healthcare Records
Brief Title: Cardiovascular Medication Use Before First Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Emily Herrett, Principle Investigator, London School of Hygiene and Tropical Medicine
Other Study IDs: CALIBER_EH3; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Antiplatelets; Lipid lowering agents; ACE inhibitors; Angiotensin Receptor Blockers; Beta blockers; Blood pressure lowering drugs
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MI patients

SUMMARY:
Large randomised trials have shown that cardiovascular medications prescribed to patients at high cardiovascular risk are effective in reducing the incidence of cardiovascular events. Their use is recommended in the United Kingdom and international guidelines (e.g. the National Institute of Clinical Excellence). However, these medications do not prevent cardiovascular events in all patients and there is now a body of research investigating the effects of cardiovascular medications on outcomes in myocardial infarction (MI), including clinical presentation, infarct size and post-MI mortality. However, the independent effects of cardiovascular drugs on post-MI all cause mortality are unclear, and there are limitations to many of the published studies in terms of their cardiovascular drug exposure data. This project utilizes prospectively collected data on cardiovascular drug use, and links to MI data from hospital and mortality records.

ELIGIBILITY:
Inclusion Criteria:

Patients in GPRD practices which are deemed "up to standard" by GPRD criteria will be included if their practice agreed to be linked to the Myocardial Ischaemic National Audit Project (MINAP), Hospital Episode Statistics (HES) and Office for National Statistics (ONS) datasets.

Patients must have at least one year of GPRD "up to standard" registration before the date of first myocardial infarction.

Age over 18. First myocardial infarction occurring between 1st January 2003 and 31st December 2008, as recorded in the HES data or MINAP.

Exclusion Criteria:

Patients will be excluded if they do not fulfil one of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients with a first myocardial infarction who are registered at those General Practice Research Database (GPRD) practices that agreed to the linkage with the MINAP database, and whose practices are "up to standard" according to GPRD criteria. Practices taking part in the GPRD are chosen to be representative of all United Kingdom (UK) practices, and 98% of people in the UK are registered with a General Practitioner (GP). Therefore the GPRD should be a representative sample of the UK population.
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Up to seven years
  All cause mortality, using Office for National Statistics (ONS) mortality statistics
Re-infarction | One year after initial myocardial infarction
  Reinfarction will be measured based on data from the General Practice Research Database (GPRD), Hospital Episode Statistics (HES), the Myocardial Ischaemia National Audit Project (MINAP) and Office for National Statistics (ONS) mortality data.

SECONDARY OUTCOMES:
Myocardial infarciton (MI) type | Measured at baseline
  Diagnosed ST-elevation MI or non ST-elevation myocardial infarction

OTHER OUTCOMES:
Infarct size | Measured at baseline
  Infarct size, as measured by levels of peak troponin in hospital, as recorded in the MINAP data source.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Herrett, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Harry Hemingway, FRCP, Study Director — University College, London
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom